CLINICAL TRIAL: NCT06356571
Title: A Single-arm, Open-label, Phase 2 Study Evaluating Subcutaneous Administration of Isatuximab, Administered by an On Body Delivery System, in Combination With Weekly Carfilzomib and Dexamethasone in Adult Participants With Relapsed and/or Refractory Multiple Myeloma (RRMM)
Brief Title: A Study to Investigate Subcutaneous Isatuximab in Combination With Weekly Carfilzomib and Dexamethasone in Adult Participants With Relapsed and/or Refractory Multiple Myeloma
Acronym: SubQSA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPS18183; U1111-1298-7348 (Other: WHO ICTRP)
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Plasma Cell Myeloma Refractory
Keywords: Anti CD38 monoclonal antibody; SARCLISA
MeSH Terms: interventions — isatuximab; montelukast; Dexamethasone; Acetaminophen; Diphenhydramine; Methylprednisolone; carfilzomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Isatuximab in combination with weekly carfilzomib and dexamethasone (Experimental): Participants will receive isatuximab via SC-OBDS administration in combination with weekly carfilzomib and dexamethasone. Isatuximab will be administered on days 1, 8, 15 and 22 for Cycle 1 and then on days 1, 15 for subsequent cycles. Carfilzomib will be administered intravenously (IV) at a starting dose on Day 1 of Cycle 1 and then escalated dose on Days 8 and 15 of Cycle 1, followed by Days 1, 8 and 15 of subsequent cycles. Dexamethasone will be given on Days 1, 8, 15, and 22 of Cycle 1 and then on Days 1, 8 and 15 of subsequent cycles. Dexamethasone will be administered IV on Cycle 1 Day 1, and IV or PO in the subsequent administrations. 1 cycle = 28 days.
  Interventions: Drug: Isatuximab SC-OBDS; Drug: Montelukast; Drug: Dexamethasone; Drug: Acetaminophen; Drug: Diphenhydramine; Drug: Methylprednisolone; Drug: Carfilzomib

INTERVENTIONS:
Drug: Isatuximab SC-OBDS — Pharmaceutical form:Solution for SC-OBDS administration-Route of administration:SC-OBDS
  Other Names: SAR650984; Sarclisa
Drug: Montelukast — Pharmaceutical form:As per local commercial product-Route of administration:Oral
Drug: Dexamethasone — Pharmaceutical form:As per local commercial product-Route of administration:Oral or IV
Drug: Acetaminophen — Pharmaceutical form:As per local commercial product-Route of administration:Oral or IV
Drug: Diphenhydramine — Pharmaceutical form:As per local commercial product-Route of administration:Oral (as premedication) or IV/oral equivalent (for management of infusion reaction)
Drug: Methylprednisolone — Pharmaceutical form:As per local commercial product-Route of administration:IV
Drug: Carfilzomib — Pharmaceutical form:As per local commercial product-Route of administration:IV

SUMMARY:
The primary purpose of this study is to assess the efficacy (overall response rate) of subcutaneous (SC) via on body delivery system (SC-OBDS) isatuximab in combination with weekly carfilzomib and dexamethasone (Kd) in adult participants with RRMM having received 1 to 3 prior lines of therapy.

DETAILED DESCRIPTION:
The duration of the study for a participant will include a period for screening of up to 28 days, a study treatment period of 12 months (except early discontinuation), the end-of-treatment (EOT) visit about 30 days after the last dose of study treatment, and a study follow-up period until death or the final study cut-off date. A cycle duration is 28 days. After study treatment discontinuation, participants will return to the study site 30 days after the last dose of study treatment for the EOT visit or before further anti-myeloma therapy initiation, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a documented diagnosis of MM.
* Participants with measurable disease defined as at least one of the following:

  * Serum M-protein ≥0.5 g/dL measured using serum protein immunoelectrophoresis and/or
  * Urine M-protein ≥200 mg/24 hours measured using urine protein immunoelectrophoresis and/or
  * Serum free light chain (FLC) assay: Involved FLC assay ≥10 mg/dL (≥100 mg/L) and an abnormal serum FLC ratio (<0.26 or >1.65).
* Participants with relapsed and/or refractory MM with at least 1 prior line of therapy and no more than 3 prior lines of therapy.
* Contraceptive use by [men and women] should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

  * Male participants agree to practice true abstinence or agree to use contraception while receiving study treatment, during dose interruptions and at least 5 months following study treatment discontinuation, even if has undergone a successful vasectomy.
  * A female participant is eligible to participate if she is not pregnant, not breastfeeding, and either is not a female of childbearing potential (FCBP XE " FCBP " \f Abbreviation \t "female of childbearing potential" ) or agrees to practice complete abstinence or use contraception.
* Capable of giving signed informed consent.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Primary refractory MM defined as participants who have never achieved at least a minimal response (MR) with any treatment during the disease course.
* Participants with prior anti-CD38 treatment if: a) administered < 6 months before first isatuximab administration or, b) intolerant to the anti-CD38 previously received.
* Participants who are refractory to carfilzomib.
* Known history of allergy to captisol (a cyclodextrin derivative used to solubilize carfilzomib), prior hypersensitivity to sucrose, histidine (as base and hydrochloride salt), polysorbate 80, or any of the components (active substance or excipient) of study treatment that are not amenable to premedication with steroids, or intolerance to arginine and Poloxamer 188 that would prohibit further treatment with these agents.
* Participants with contraindication to dexamethasone and/or to carfilzomib.
* Any anti-myeloma drug treatment within 14 days before the first isatuximab administration, including dexamethasone.
* Prior allogenic HSC transplant with active graft versus host disease (GvHD XE " GvHD " \f Abbreviation \t "graft versus host disease" ) (GvHD any grade and/or being under immunosuppressive treatment within the last 2 months).
* Any major procedure within 14 days before the first isatuximab administration: plasmapheresis, major surgery (kyphoplasty is not considered a major procedure), radiotherapy.
* Vaccination with a live vaccine within 4 weeks before the first isatuximab administration. Seasonal flu vaccines that do not contain live virus are permitted.
* Participant not suitable for participation, whatever the reason, as judged by the Investigator, including medical or clinical conditions, or participants potentially at risk of noncompliance to study procedures.

The above information is not intended to contain all considerations relevant to the potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2027-01-08 (Estimated); Study Completion 2027-07-15 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 6 months after the Last Participant In (LPI) i.e., approximately 32 months
  ORR, defined as the proportion of participants with stringent complete response (sCR), complete response (CR), very good partial response (VGPR), and partial response (PR), according to IMWG criteria assessed by investigator.

SECONDARY OUTCOMES:
Number of participants with infusion reactions (IRs) | From the signing of informed consent to 30 days after the date of the last study treatment administration i.e., approximately 38 months
Number of participants with treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), and laboratory abnormalities (per NCI-CTCAE grade or PCSA if NCI-CTCAE scale is not applicable) | From the signing of informed consent to 30 days after the date of the last study treatment administration i.e., approximately 38 months
Number of participants with injection site reactions (ISRs) | From the signing of informed consent to 30 days after the date of the last study treatment administration i.e., approximately 38 months
CR or better | 12 months after the Last Participant In (LPI) i.e., approximately 38 months
  CR or better assessed according to International Myeloma Working Group (IMWG) criteria assessed by investigator. CR is defined as negative immunofixation on the serum and urine, and disappearance of any soft tissue plasmacytomas, <5% plasma cells in bone marrow aspirates, and a normal FLC ratio of 0.26-1.65 is required for FLC disease only. Two consecutive assessments are needed. No known evidence of progressive disease or new bone/soft tissue lesions if radiographic studies were performed.
VGPR or better | 12 months after the Last Participant In (LPI) i.e., approximately 38 months
  VGPR or better assessed according to IMWG criteria assessed by investigator. VGPR is defined as Serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥90% reduction in serum M-protein plus urine M-protein level <100 mg/24 h, or ≥90% decrease in the sum of maximal perpendicular diameter compared to baseline in soft tissue plasmacytoma. FLC only: a ≥90% decrease in the difference between involved and uninvolved FLC levels. Two consecutive assessments are needed. No known evidence of progressive disease or new bone/soft tissue lesions if radiographic studies were performed.
Duration of response (DOR) | 12 months after the Last Participant In (LPI) i.e., approximately 38 months
  DOR, defined as the time from date of first investigator determined response for achieving PR or better to first documentation of progressive disease (PD) determined by investigator or death, whichever occurred first.
Time to first response (TT1R) | 12 months after the Last Participant In (LPI) i.e., approximately 38 months
  TT1R, defined as the time from first isatuximab administration to first investigator-determined response (PR or better) that is subsequently confirmed.
Time to best response (TTBR) | 12 months after the Last Participant In (LPI) i.e., approximately 38 months
  TTBR, defined as the time from first isatuximab administration to first occurrence of investigator-determined best response (PR or better) that is subsequently confirmed.
Patient experience and Satisfaction Questionnaire v2 (PESQ v2) | Cycle 3/Day 15 and Cycle 6/Day 15
  The PESQ v2 has been designed to follow up on participant experience and satisfaction regarding the treatment (side effects and recommendation) and the administration method (comfortability, pain, side effects and overall satisfaction). This questionnaire has been developed using industry standard for instrument development and has been debriefed and adapted based on qualitative interviews with oncology patients. The more general treatment expectations instrument (v1) was further adapted and debriefed with patients to assess manual and OBDS subcutaneous delivery (v2). The trial specific version of the PESQ v2 contains of items administered for the duration of treatment. Response options are presented as a 5-point Likert scale ranging from Strongly agree/very satisfied/definitely yes to strongly disagree/very dissatisfied/definitely no.
Positivity titer of anti-drug antibodies (ADA) in a subset of approximately 30 participants | From Cycle 1 Day 1 to follow-up (90 days from last administration) i.e, approximately up to 15 months (1 cycle = 28 days)
  Blood samples will be collected for assessing the presence of ADA against isatuximab in plasma from approximately 30 participants. Plasma samples will be screened for antibodies binding to isatuximab and the titer of confirmed positive samples will be reported.
Maximum observed concentration (Cmax) of isatuximab in a subset of approximately 30 participants | Multiple timepoints in Cycle 1 (1 cycle = 28 days)
Cumulative area under the curve over the first 4 weeks of isatuximab treatment (AUC4 weeks) in a subset of approximately 30 participants | Multiple timepoints in Cycle 1 (1 cycle = 28 days)

CONTACTS AND LOCATIONS:
Locations (31):
- United States (31):
  - Mayo Clinic in Arizona - Phoenix- Site Number : 8400058, Phoenix, Arizona
  - Private Practice - Dr. James R. Berenson- Site Number : 8400044, West Hollywood, California
  - Smilow Cancer Center at Yale-New Haven- Site Number : 8400020, New Haven, Connecticut
  - Maryland Oncology Hematology- Site Number : 8400038, Washington D.C., District of Columbia
  - Center for Rheumatology, Immunology and Arthritis- Site Number : 8400031, Fort Lauderdale, Florida
  - Mayo Clinic in Florida- Site Number : 8400002, Jacksonville, Florida
  - Florida Cancer Specialists- Site Number : 8400030, Lake Mary, Florida
  - The Oncology Institute of Hope & Innovation - Lakeland- Site Number : 8400054, Lakeland, Florida
  - D&H Pompano Research Center- Site Number : 8400049, Margate, Florida
  - Millennium Oncology - Pembroke Pines- Site Number : 8400011, Pembroke Pines, Florida
  - BRCR Global- Site Number : 8400008, Plantation, Florida
  - Pontchartrain Cancer Center - Covington- Site Number : 8400046, Covington, Louisiana
  - Beth Israel Deaconess Medical Center - Boston- Site Number : 8400005, Boston, Massachusetts
  - Michigan Hematology & Oncology Consultants - Dearborn- Site Number : 8400036, Dearborn, Michigan
  - Hematology Oncology Consultants - Royal Oak- Site Number : 8400039, Royal Oak, Michigan
  - Alliance for Multispeciality Research - Kansas City- Site Number : 8400056, Kansas City, Missouri
  - Washington University- Site Number : 8400007, St Louis, Missouri
  - Hackensack Meridian Health - Hackensack University Medical Center- Site Number : 8400021, Hackensack, New Jersey
  - San Juan Oncology Associates- Site Number : 8400016, Farmington, New Mexico
  - Memorial Sloan Kettering Cancer Center - New York - York Avenue- Site Number : 8400003, New York, New York
  - Duke University Medical Center- Site Number : 8400018, Durham, North Carolina
  - Gabrail Cancer Center- Site Number : 8400010, Canton, Ohio
  - University of Cincinnati Medical Center- Site Number : 8400043, Cincinnati, Ohio
  - Oncology Hematology Care - Kenwood- Site Number : 8400014, Cincinnati, Ohio
  - Roper Saint Francis Healthcare- Site Number : 8400013, Charleston, South Carolina
  - Prisma Health Cancer Institute - Greenville- Site Number : 8400019, Greenville, South Carolina
  - Gibbs Cancer Center-Spartanburg Medical Center- Site Number : 8400001, Spartanburg, South Carolina
  - Tennessee Cancer Specialists - Knoxville - Old Weisgarber Road- Site Number : 8400035, Knoxville, Tennessee
  - University of Tennessee Medical Center- Site Number : 8400006, Knoxville, Tennessee
  - Virginia Cancer Specialists- Site Number : 8400045, Fairfax, Virginia
  - SSM Health Dean Medical Group - Wisconsin - Madison- Site Number : 8400009, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: LPS18183 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25728&tenant=MT_SNY_9011